CLINICAL TRIAL: NCT00219648
Title: A Phase II, Randomized, Double-Blind, Placebo-Controlled, Parallel Group, Dose- Finding, Two-Stage Study to Assess the Efficacy and Safety of 12 Weeks of Treatment With PEP03 in Patients With Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: Two-Stage Study to Assess the Efficacy and Safety of 12 Weeks of Treatment With PEP03 in Patients With Chronic Obstructive Pulmonary Disease (COPD)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: PharmaEngine (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PEP0301
Record Dates: First submitted 2005-09-20; First posted 2005-09-22 (Estimated); Last update posted 2005-09-22 (Estimated); Status verified 2005-09

CONDITIONS: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

INTERVENTIONS:
Drug: PEP03

SUMMARY:
PEP03 is a new chemical entity developed as a highly selective, potent, and orally active 5-LO inhibitor. PEP03 exerts its action by blocking the generation of both cysteinyl LTs and LTB4. These LTs have been associated with the inflammatory response in the lung and with the clinical sequelae, including bronchospasm. Preclinical pharmacological in- vitro, ex-vivo and in-vivo testing indicates that PEP03 has multiple beneficial actions including prevention of bronchoconstriction, and reduction of vascular leakage, cellular infiltration, and bronchial hyperresponsiveness.

Clinical studies in asthmatic patients indicate that PEP03 improved FEV1 and other secondary endpoints, such as morning and evening peak flow, daytime and nighttime symptoms score, beta-agonist use, physician's and patient's global impression of change. Since leukotrienes have been suggested to be involved in the pathophysiology of COPD, this study is designed to explore the clinical utility of PEP03 for the treatment of moderate COPD.6; 7; 8; 9

ELIGIBILITY:
Inclusion Criteria:

* 1. Subjects have to be > 40 years of age. 2. Subjects must have baseline 40% ≦ FEV1(pre-bronchodilator) ≦ 70% of predicted value, and FEV1/FVC < 70% at Visits 1 and 2.

  3. Subjects must have at least one episode of COPD-related symptoms (e.g. cough, sputum production, shortness of breath) within 2 months prior to screening.

  4. Subjects must have a < 12% increase in FEV1 after a fixed dose of bronchodilator (200 g inhaled salbutamol).

  5. Subjects have a history of > 10 pack years of smoking (1 pack year = 20 cigarettes smoked per day for 1 year or equivalent).

  6. Subjects of childbearing potential must use adequate birth control measures and must have a negative serum pregnancy test prior to study entry.

  7. Subjects have to be able to adhere to the study visit schedule and other protocol requirements.

  8. Subjects must have the ability to use peak flow meter correctly and record patient diary cards 9. Subjects must provide signed, written informed consent prior to participation in the study.

Exclusion Criteria:

* 1. Subjects have asthma, allergic rhinitis or atopy as main component of their obstructive airway disease.

  2. Subjects are being treated with long term oxygen therapy, requiring supplemental oxygen more often than on an occasional/as need basis or requiring nocturnal positive pressure for sleep apnea.

  3. Subjects have a history of severe right sided heart failure or cor pulmonale.

  4. Subjects have had a serious infection (e.g. hepatitis, pneumonia or pyelonephritis) within the previous 3 months.

  5. Subjects have airway obstruction due to diseases with known etiology or specific pathology, such as cystic fibrosis, or bronchiectasis.

  6. Subjects with lung cancer, sarcoidosis, tuberculosis, or lung fibrosis. 7. Subjects with a history of drug or alcohol abuse. 8. Subjects have used investigational drugs within 1 month prior to screening or within 5 half-lives of the investigational agent, whichever is longer.

  9. Subjects are currently treated with cromolyn sodium or nedocromil, long-acting theophylline, leukotriene modifiers, oral or inhaled corticosteroids, long acting β2-agonists, or long-acting anticholinergics.

  10. Subjects with liver enzymes (AST, ALT, bilirubin) > 3 X upper limit of normal range.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2004-09

CONTACTS AND LOCATIONS:
Locations (1):
- Chang Gung Memorial Hospital, Taipei, Taiwan